CLINICAL TRIAL: NCT05545787
Title: A Prospective, Randomized, Non-inferiority Study to Compare Efficacy and Safety of Cold Snare Endoscopic Mucosal Resection and Hot Snare Endoscopic Mucosal Resection in Treatment for 10-19 mm Non-pedunculated Colorectal Polyps
Brief Title: Cold or Hot Snare Endoscopic Mucosal Resection for 10-19mm Non-pedunculated Colorectal Polyps
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qingwei Jiang (Other)
Responsible Party: Sponsor-Investigator, Qingwei Jiang, attending physician, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K2203
Record Dates: First submitted 2022-09-15; First posted 2022-09-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Polyp

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cold snare endoscopic mucosal resection (CS-EMR) (Experimental): Eligible colorectal polyps sized 10-19mm will be resected by CS-EMR
  Interventions: Procedure: Cold snare endoscopic mucosal resection
- Hot snare endoscopic mucosal resection (HS-EMR) (Experimental): Eligible colorectal polyps sized 10-19mm will be resected by HS-EMR
  Interventions: Procedure: Hot snare endoscopic mucosal resection

INTERVENTIONS:
Procedure: Cold snare endoscopic mucosal resection — During CS-EMR, methylene blue-tinted epinephrine saline will be injected into the submucosal space around the lesion to lift the lesion. The polyp and 1-2mm of surrounding mucosa will then be closely snared and transected mechanically.
  Arms: Cold snare endoscopic mucosal resection (CS-EMR)
Procedure: Hot snare endoscopic mucosal resection — During HS-EMR, methylene blue-tinted epinephrine saline will be injected into the submucosal space around the lesion to lift the lesion. The snare will be placed around the lesion, and then cautery will be applied using the electrosurgical generator.
  Arms: Hot snare endoscopic mucosal resection (HS-EMR)

SUMMARY:
This is a prospective, randomized, open-label, non-inferiority, multiple-center trial. Outpatients who are scheduled to undergo colonoscopy and found eligible polyps will be randomized to receive either cold snare endoscopic mucosal resection (CS-EMR) or hot snare endoscopic mucosal resection (HS-EMR). This study aims to compare the efficacy and safety of CS-EMR or HS-EMR for the resection of non-pedunculated colorectal polyps sized 10-19mm.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age;
* undergo colonoscopy in the Digestive Endoscopy Center of Peking Union Medical College Hospital, Beijing Tsinghua Changgung Hospital or Seventh Medical Center, General Hospital of the Chinese People's Liberation Army;
* volunteer to participate in this study and sign informed consent;
* at least one polyp sized 10-19 mm (Paris classification Is or IIa) by colonoscopy.

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) status class 3 or above;
* poor bowel preparation (Boston bowel preparation scale < 6 points);
* known or endoscopic features indicating the submucous infiltration or malignancy;
* oral anti-coagulants, or antiplatelet agents, or known blood coagulation disorders, or bleeding tendency (platelets<50000 cells/mm3 or INR>1.5);
* a history of colorectal resection;
* emergency colonoscopy (hemodynamic instability and/or continued active gastrointestinal bleeding and/or requiring intensive care patients);
* inflammatory bowel disease, familial polyposis, and colorectal cancer;
* pregnancy or lactation;
* severe cardiopulmonary dysfunction, liver cirrhosis, chronic kidney disease, other malignant tumors, or severe infectious diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Complete resection rate | Within 14 days
  The resection is considered histologically complete if the lateral margins of the resected polyps are surrounded by normal tissue and the vertical margin is free of neoplasia tissue. If en-bloc resection is not achieved, 5 biopsies (4 biopsies obtained in a 4-quadrant fashion from the polypectomy site margins; 1 biopsy from the base) are applied to evaluate histological completeness of resection.

SECONDARY OUTCOMES:
En-bloc resection rate | Within 1 day
  The lesion was completely excised under endoscope and a single specimen was obtained.
Intraprocedural bleeding | Within 1 day
  Any immediate episode requiring any form of endoscopic hemostasis or oozing for more than 60s
Intraprocedural perforation | Within 1 day
  Endoscopic observation of perforation requiring sealing with clips
Delayed bleeding | Within 14 days
  Any episode requiring emergency department presentation, hospitalization, or reintervention within 14 days
Delayed perforation | Within 14 days
  Any perforation within 14 days
Number of clips used | Within 1 day
  The number of endoscopic clips used for each resected polyp
Resection time | Within 1 day
  The duration from the first occurrence of injection needle under endoscope visual field to complete removal of the resected polyp
Total cost | Within 1 day
  Total cost including both treatment cost and material cost for polyp resection

CONTACTS AND LOCATIONS:
Overall Officials: Qingwei Jiang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (14):
- China (14):
  - Beijing Dongcheng District First People's Hospital, Beijing, Beijing Municipality
  - Emergency General Hospital, Beijing, Beijing Municipality
  - Beijing Sixth Hospital, Beijing, Beijing Municipality
  - Seventh Medical Center, General Hospital of the Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Beijing Fangshan District Liangxiang Hospital, Beijing, Beijing Municipality
  - Beijing Daxing District People's Hospital, Beijing, Beijing Municipality
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Longquan Hospital, Sichuan University, Chengdu, Sichuan
  - PLA Western Theater General Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang Q, Yan X, Wang D, Zhang S, Zhang Y, Feng Y, Yang A, Wu D. Endoscopic mucosal resection using cold snare versus hot snare in treatment for 10-19 mm non-pedunculated colorectal polyps: protocol of a non-inferiority randomised controlled study. BMJ Open. 2023 May 22;13(5):e070321. doi: 10.1136/bmjopen-2022-070321. PMID 37217262